CLINICAL TRIAL: NCT01821430
Title: Opioid-Induced Hyperalgesia in Prescription Opioid Abusers: Effects of Pregabalin
Brief Title: Increased Sensitivity to Pain Caused by Opioids in People Who Have Abused Prescription Opioids
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: poor recruitment
Sponsor: Georgetown University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Peggy Compton, Professor and Associate Dean, Georgetown University
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00000669; U01DA029580 (NIH)
Record Dates: First submitted 2013-03-27; First posted 2013-04-01 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2017-02

CONDITIONS: Chronic Pain
Keywords: Chronic Pain; Narcotic Abuse; Opioid related disorders; Opiate substitution treatment; Buprenorphrine; Pregabalin; Methadone
MeSH Terms: conditions — Chronic Pain; Narcotic-Related Disorders; Opioid-Related Disorders | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pregabalin (Experimental): Pregabalin 400mg / Day
  Interventions: Drug: Pregabalin
- Placebo Control (Placebo Comparator): Placebo Tablet
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pregabalin — Titration of intervention will begin with 50mg PO BID x 2 days, then 100mg PO BID x 2 days, then 150mg PO BID X 2 days, then on day 7 full dose of Pregabalin 400mg PO QD for six weeks
  Other Names: Lyrica
  Arms: Pregabalin
Drug: Placebo — Placebo group will follow the same titration as the pregabalin group
  Arms: Placebo Control

SUMMARY:
Managing pain in patients who abuse prescription opioids presents many challenges, including the development of opioid-induced hyperalgesia (OIH). Hyperalgesia is a condition in which something that usually feels slightly painful is perceived as something very painful. The proposed study will test the efficacy of the well-known neurological medication pregabalin to diminish OIH and chronic pain in persons who are in Suboxone (buprenorphine) or methadone treatment for prescription drug abuse.

DETAILED DESCRIPTION:
The clinical management of pain in prescription opioid abusers presents a challenge to the health care professional. Investigators have novel pilot data showing that the GABA-agonist gabapentin (GPN) significantly decreases opioid-induced hyperalgesia (OIH) in methadone patients (Compton et al., 2009), providing the first empirical evidence of a pharmacotherapy for OIH in opioid abusers. The work of Gore and colleagues (2011) showed that pregabalin (PGB), a GABA analogue succeeding GPN, was shown to decrease opioid use in patients with neuropathic pain in patients, suggesting an anti-hyperalgesia effect not observed in the matched cohort receiving GPN. The proposed research will comprehensively evaluate the efficacy of PGB in treating opioid-induced hyperalgesia (OIH) in a well-described population of prescription opioid abusers (POAs) with chronic pain and on Suboxone (buprenorphine) or methadone therapy. A pressing need for such investigation is presented by the rising number of POAs presenting for treatment (SAMHSA, 2010; 2011), and for whom, chronic pain is a common co-morbidity. The proposed work is anticipated to provide vital and timely information on the efficacy of PGB in the treatment of OIH in prescription opioid abusers on Suboxone or methadone therapy.

Following recruitment and screening, 75 subjects assigned to the active medication group will receive pregabalin 400 mg/day, a dose well-within published guidelines of 300-600 mg/day for the treatment of neuropathic pain (http://www.pfizerpro.com/hcp/lyrica/phndosing). During the first week of treatment, subjects will be quickly titrated up to the assigned daily PGB dose of 400 mg/day PO (50mg BID x 2 days; 100mg BID x 2 days; 150mg BID x 2 days, with full dosage of 400mg administered on day 7 ), or maximum dose tolerated) for six weeks. 75 subjects will be assigned to receive matched and undergo identical titration and study activities under double-blind conditions. Study staff will evaluate subjects daily by phone during titration; thereafter they will be seen weekly at study sessions. Tapering of medication will begin at the end of week 6. The severity of chronic pain will be measured at each time point using two standardized self report tools which report on pain severity (McGill Pain Questionnaire) and pain-related disability (Brief Pain Inventory). Opioid-induced hyperalgesia will be measured at each time point using a standardized cold pressor trial, and performance at baseline will be compared to performance following PGB/placebo administration over time.

ELIGIBILITY:
Inclusion Criteria:

1. Be between the ages of 21 and 65 years of age.
2. Have a DSM-IVR diagnosis (used through 10/1/2014) of prescription opioid abuse or dependence disorder or a DSM-5 diagnosis of opioid use disorder.
3. Be enrolled and compliant in Suboxone or methadone treatment and on a stable dose [Suboxone (6-24mg/day); of methadone (60-120mg/day)] x at least 10 days.
4. Provide urine sample absent of any non-prescribed drugs of abuse at screening.
5. Screening cold-pressor pain tolerance < 70 seconds
6. Have chronic lower back pain or arthritis pain (duration six or more months).
7. Be otherwise in good physical health, or in the case of a medical condition needing ongoing treatment, be in the care of a physician who is willing to take responsibility for such treatment. The same conditions apply in cases of patients with a psychiatric disorder needing ongoing treatment.
8. Be agreeable to and capable of signing an informed consent.

Exclusion Criteria:

1. Have known sensitivity to pregabalin or gabapentin.
2. Potential participants must not be taking the following medications: pregabalin or gabapentin, tiagabine, vigabatrin, valproate, phenobarbital or primidone for the treatment of epilepsy; SNRI or TCA antidepressants; baclofen; or carbamazepine, oxycarbazepine or lamotrigine for the treatment of chronic pain.
3. Currently be substance dependent on alcohol, benzodiazepine, methamphetamine, cocaine or other drugs of abuse (except nicotine).
4. Have any acute medical condition that would make participation medically hazardous, (e.g., acute hepatitis, unstable cardiovascular disease, liver or renal disease) or have liver enzyme values (AST or ALT) greater than 5 times normal range.
5. Be acutely psychotic, severely depressed and in need of inpatient treatment, or an immediate suicide risk.
6. Have a neurological or psychiatric illness (i.e., schizophrenia, Raynaud's disease, urticaria, stroke) that would affect pain responses.
7. Be currently taking opioid analgesic medication for a painful condition on a regular basis.
8. Be a nursing or pregnant female, or a female or male who does not agree to not become pregnant or father a child during the course of, and six months following completion of the study. If a subject becomes pregnant or fathers a child during the study, they must immediately notify the study investigator.
9. Have a history of heart disease, stroke, liver or kidney disease, epilepsy or acute hepatitis, or currently have a pacemaker or uncontrolled high blood pressure.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Improved Pain Response, threshold and tolerance | 8 weeks
  To test the efficacy of PGB, compared to placebo, to diminish OIH, as evidenced by improved pain responses (threshold and tolerance) to experimentally induced cold-pressor pain, in a well-described sample of POA patients with chronic pain and on buprenorphine or methadone therapy.
  * Pain Threshold: On the CP assay, pain threshold is operationalized as the number of seconds after the onset of the painful stimulus when a painful sensation is first detected. Subjects will indicate threshold by saying "Pain."
  * Pain Tolerance: On the CP assay, pain tolerance is operationalized as the number of seconds after the onset of the painful stimulus when the painful sensation is subjectively intolerable. Subjects will indicate tolerance by removing their arm from the ice bath.

SECONDARY OUTCOMES:
Improvement in pain severity and daily functionality | 8 weeks
  To test the efficacy of PGB, compared to placebo, to diminish chronic pain, as evidenced by improvements in pain severity and functionality in a well-described sample of POA patients with chronic pain and on buprenorphine or methadone therapy.
  Pain Severity will be measured with The McGill Pain Questionnaire. Daily Functionality will be measured with the Brief Pain Inventory

CONTACTS AND LOCATIONS:
Overall Officials: Peggy Compton, RN, PhD, Principal Investigator — Georgetown University
Locations (1):
- Georgetown University, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Backonja MM. Anticonvulsants (antineuropathics) for neuropathic pain syndromes. Clin J Pain. 2000 Jun;16(2 Suppl):S67-72. doi: 10.1097/00002508-200006001-00012. PMID 10870743
- [Background] Barrett AC, Smith ES, Picker MJ. Capsaicin-induced hyperalgesia and mu-opioid-induced antihyperalgesia in male and female Fischer 344 rats. J Pharmacol Exp Ther. 2003 Oct;307(1):237-45. doi: 10.1124/jpet.103.054478. Epub 2003 Sep 3. PMID 12954802
- [Background] Ben-Menachem E. Pregabalin pharmacology and its relevance to clinical practice. Epilepsia. 2004;45 Suppl 6:13-8. doi: 10.1111/j.0013-9580.2004.455003.x. PMID 15315511
- [Background] Blitz B, Dinnerstein AJ, Lowenthal M. Performance on the pain apperception test and tolerance for experimental pain: a lack of relationship. J Clin Psychol. 1968 Jan;24(1):73. doi: 10.1002/1097-4679(196801)24:13.0.co;2-5. No abstract available. PMID 4867371
- [Background] Chen ACN, Dworkin SF, Haug J, Gehrig J. Human pain responsivity in a tonic pain model: psychological determinants. Pain. 1989 May;37(2):143-160. doi: 10.1016/0304-3959(89)90126-7. PMID 2664663
- [Background] Chery-Croze S. Relationship between noxious cold stimuli and the magnitude of pain sensation in man. Pain. 1983 Mar;15(3):265-9. doi: 10.1016/0304-3959(83)90061-1. PMID 6856323
- [Background] Cleeland CS, Ryan KM. Pain assessment: global use of the Brief Pain Inventory. Ann Acad Med Singap. 1994 Mar;23(2):129-38. PMID 8080219
- [Background] Compton P, Charuvastra VC, Ling W. Pain intolerance in opioid-maintained former opiate addicts: effect of long-acting maintenance agent. Drug Alcohol Depend. 2001 Jul 1;63(2):139-46. doi: 10.1016/s0376-8716(00)00200-3. PMID 11376918
- [Background] Compton PA, Ling W, Torrington MA. Lack of effect of chronic dextromethorphan on experimental pain tolerance in methadone-maintained patients. Addict Biol. 2008 Sep;13(3-4):393-402. doi: 10.1111/j.1369-1600.2008.00112.x. Epub 2008 May 26. PMID 18507735
- [Background] Compton P, Kehoe P, Sinha K, Torrington MA, Ling W. Gabapentin improves cold-pressor pain responses in methadone-maintained patients. Drug Alcohol Depend. 2010 Jun 1;109(1-3):213-9. doi: 10.1016/j.drugalcdep.2010.01.006. Epub 2010 Feb 16. PMID 20163921
- [Background] Gore M, Tai KS, Zlateva G, Bala Chandran A, Leslie D. Clinical characteristics, pharmacotherapy, and healthcare resource use among patients with diabetic neuropathy newly prescribed pregabalin or gabapentin. Pain Pract. 2011 Nov-Dec;11(6):528-39. doi: 10.1111/j.1533-2500.2011.00450.x. Epub 2011 Mar 16. PMID 21435162
- [Background] Hansen GR. The drug-seeking patient in the emergency room. Emerg Med Clin North Am. 2005 May;23(2):349-65. doi: 10.1016/j.emc.2004.12.006. PMID 15829387
- [Background] Holtman JR Jr, Wala EP. Characterization of the antinociceptive and pronociceptive effects of methadone in rats. Anesthesiology. 2007 Mar;106(3):563-71. doi: 10.1097/00000542-200703000-00022. PMID 17325516
- [Background] Ifuku M, Iseki M, Hidaka I, Morita Y, Komatus S, Inada E. Replacement of gabapentin with pregabalin in postherpetic neuralgia therapy. Pain Med. 2011 Jul;12(7):1112-6. doi: 10.1111/j.1526-4637.2011.01162.x. Epub 2011 Jun 21. PMID 21692969
- [Background] Paulson MR, Dekker AH, Aguilar-Gaxiola S. Eliminating disparities in pain management. J Am Osteopath Assoc. 2007 Sep;107(9 Suppl 5):ES17-20. PMID 17908826
- [Background] Ramanujam VM, Anderson KE, Grady JJ, Nayeem F, Lu LJ. Riboflavin as an oral tracer for monitoring compliance in clinical research. Open Biomark J. 2011;2011(4):1-7. doi: 10.2174/1875318301104010001. PMID 21949554
- [Background] Tassone DM, Boyce E, Guyer J, Nuzum D. Pregabalin: a novel gamma-aminobutyric acid analogue in the treatment of neuropathic pain, partial-onset seizures, and anxiety disorders. Clin Ther. 2007 Jan;29(1):26-48. doi: 10.1016/j.clinthera.2007.01.013. PMID 17379045
- [Background] Tassorelli C, Micieli G, Osipova V, Rossi F, Nappi G. Pupillary and cardiovascular responses to the cold-pressor test. J Auton Nerv Syst. 1995 Oct 5;55(1-2):45-9. doi: 10.1016/0165-1838(95)00026-t. PMID 8690850
- [Background] Bodian D. Origin of specific synaptic types in the motoneuron neuropil of the monkey. J Comp Neurol. 1975 Jan 15;159(2):225-43. doi: 10.1002/cne.901590205. PMID 1112912